CLINICAL TRIAL: NCT00288561
Title: Open-Label, Multicenter, Phase II Study Assessing the Safety of Ranibizumab Administered in Conjunction With Photodynamic Therapy With Verteporfin in Patients With Occult or Predominately Classic Subfoveal Choroidal Neovascularization (CNV) Secondary to Age-Related Macular Degeneration (ARMD)
Brief Title: Study of Ranibizumab Administered in Conjunction With Photodynamic Therapy With Verteporfin in Patients With Subfoveal Choroidal Neovascularization and Age-Related Macular Degeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002B2201
Record Dates: First submitted 2006-02-07; First posted 2006-02-08 (Estimated); Last update posted 2008-06-19 (Estimated); Status verified 2008-06

CONDITIONS: Age-Related Macular Degeneration (ARMD)
Keywords: ARMD, ranibizumab, verteporfin
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

INTERVENTIONS:
Drug: ranibizumab

SUMMARY:
Ranibizumab is derived from a murine monoclonal anti- vascular endothelial growth factor (VEGF) antibody and can penetrate through the many retinal cell layers following intravitreal injection. The present study is directed towards the assessment of ranibizumab administered on the same day in combination with verteporfin in patients with subfoveal CNV secondary to ARMD

ELIGIBILITY:
Inclusion Criteria:

* Patients 50 years of age or greater who have provided written informed consent

  * Patients with subfoveal choroidal neovascularization lesions secondary to AMD, either predominantly classic or occult with no classic component
  * Patients who have a BCVA score between 73 and 24 letters, inclusively, in the study eye using ETDRS (approximately 20/40 to 20/320)
  * Willing to return for all scheduled visits

Exclusion Criteria:

* - Patients who have a BCVA of < 34 letters in both eyes (legally blind is defined as bilateral vision below 20/200 or less than 34 letters)
* Prior treatment in the study eye with verteporfin, external-beam radiation therapy, subfoveal focal laser photocoagulation, vitrectomy, or transpupillary thermotherapy
* Previous participation in a clinical trial (for either eye) involving anti-angiogenic drugs (pegaptanib, ranibizumab, anecortave acetate, protein kinase C inhibitors, etc.)

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-11; Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Customer Information, Study Chair — Novartis - Including Sites in Germany
Locations (1):
- Novartis, Basel, Switzerland